CLINICAL TRIAL: NCT01373658
Title: Safety and Efficacy Registry of Yinyi Polymer-free Paclitaxel-eluting Stent
Brief Title: Safety and Efficacy Registry of Yinyi Stent (SERY-II)
Acronym: SERY-II
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Weifeng Shen, Ruijin hospital, shanghai jiao tong university school of medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH20100910
Record Dates: First submitted 2011-04-01; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yinyi stent (Experimental)
  Interventions: Device: Yinyi stent

INTERVENTIONS:
Device: Yinyi stent — subjects with Yinyi stent implantation

SUMMARY:
Drug-eluting stents effectively reduce restenosis but may increase late thrombosis and delayed restenosis. Persistent polymer could be responsible. Local delivery of paclitxel from a polymer-free Yinyi stent (Dalian Yinyi biomaterial research and development co.ltd) may prevent these complications.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* both gender
* native coronary lesion
* narrowing > 70%
* vessel size 2.5-4.0 in diameter

Exclusion Criteria:

* without informed consent,
* ST elevation myocardial infarction within 7 days,
* patient with ≤ 70% coronary narrowing at target lesion,
* left main lesion,
* multivessel narrowing need more than 3 stent implantations,
* by-pass graft,
* abnormal liver function before randomization,
* active hepatitis or muscular disease,
* impaired renal function with serum creatinine level > 3mg/dl,
* impaired left ventricular function with LVEF < 30%,
* participate in other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
late lumen loss | 12 months
  Late luminal loss was defined as the difference between the minimal luminal diameter immediately after the placement of the stent and the minimal luminal diameter at 12-month angiographic follow-up.

SECONDARY OUTCOMES:
major adverse cardiac events | 12 months
  including cardiac death, re-infarction, and target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- ruijin hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China